CLINICAL TRIAL: NCT01031498
Title: Phase II, Open, Randomized Comparative Trial of Two Different Schedules of Palonosetron Versus Ondansetron for the Prevention of Nausea and Vomiting in Patients With Hematologic Malignancies Receiving Regimens Containing High-dose Cytarabine
Brief Title: Palonosetron Versus Ondansetron for the Prevention of Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0389
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myelogenous Leukemia; Chemotherapy-induced Nausea and Vomiting
Keywords: Nausea; Vomiting; CINV; Leukemia; High-risk Myelodysplastic syndrome; AML; Hematologic malignancies; Hematologic Disorder; Continuous multi-day chemotherapy; High-dose cytarabine; Palonosetron; Aloxi; Ondansetron; Zofran
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Vomiting; Nausea; Leukemia; Hematologic Neoplasms; Hematologic Diseases | interventions — Ondansetron; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ondansetron: Standard of Care (Active Comparator): Standard of care, Ondansetron 8 mg IV as bolus followed by 24 mg IV from 30 minutes before chemotherapy until 12 hours after chemotherapy ends.
  Interventions: Drug: Ondansetron
- Palonosetron Group 1 (5 Days) (Experimental): Palonosetron once a day 0.25 mg IV injection for 5 days, given over 30 seconds, 30 minutes before chemotherapy treatment.
  Interventions: Drug: Palonosetron
- Palonosetron Group 2 (3 Days) (Experimental): Palonosetron once a day 0.25 mg IV injection on Days 1, 3, and 5 of chemotherapy treatment, given over 30 seconds, 30 minutes before chemotherapy treatment.
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Ondansetron — 8 mg IV as bolus followed by 24 mg IV from 30 minutes before chemotherapy until 12 hours after chemotherapy ends.
  Other Names: Zofran
  Arms: Ondansetron: Standard of Care
Drug: Palonosetron — Palonosetron Group 1: 0.25 mg IV bolus over 30 seconds daily for 5 days, 30 minutes before cytarabine chemotherapy.
  Palonosetron Group 2: 0.25 mg IV bolus over 30 seconds on Days 1, 3, and 5 of cytarabine chemotherapy, 30 minutes before chemotherapy.
  Other Names: Aloxi
  Arms: Palonosetron Group 1 (5 Days); Palonosetron Group 2 (3 Days)

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of 3 drug schedules in preventing chemotherapy-related nausea and/or vomiting in patients with acute myelogenous leukemia (AML) or high-risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Chemotherapy-related nausea and vomiting is a frequent problem among patients with leukemia that can lead to further medical problems, such as malnutrition, dehydration, electrolyte imbalance, and a lower quality of life. Cytarabine, one of the drugs that is used to treat AML and high-risk MDS, is known to cause nausea and/or vomiting, so all patients that receive chemotherapy with cytarabine also need to receive medication to prevent these side effects.

One standard-of-care drug to treat chemotherapy-related nausea and vomiting is called Ondansetron. Palonosetron is a new drug similar to Ondansetron that is designed to stay longer in the bloodstream. Researchers want to find out if palonosetron can prevent nausea and vomiting better than ondansetron.

Women who are able to have children must have a negative blood or urine pregnancy test before starting treatment.

If you are still eligible to take part in this study, you will be randomly assigned (as in the roll of the dice) to one of 3 treatment groups. Participants in the first group will be given Ondansetron as an intravenous (IV--through a needle in your vein) continuous infusion, from 30 minutes before your chemotherapy treatment until 12 hours after chemotherapy ends. This is considered the standard of care.

Participants assigned to the second treatment group will be given palonosetron once a day by IV injection for 5 days. Each dose will be given over a period of 30 seconds, 30 minutes before your chemotherapy treatment.

Participants assigned to the third treatment group will be given palonosetron once a day by IV injection, on Days 1, 3, and 5 of chemotherapy treatment. Each dose will be given over a period of 30 seconds, 30 minutes before your chemotherapy treatment.

No matter what group you are assigned to, you will receive extra medication for nausea and/or vomiting as needed.

You will be asked to fill out a study diary daily for 7 days, and it should take you no longer than 10 minutes to complete. The diary will be used to record the number of episodes of nausea and/or vomiting you experience during this study, as well as to record any need for extra medications, and to help researchers learn which of the 2 drugs helps the best to improve participants' quality of life (such as sleep, daily activities, and your ability to think and reason).

You will be taken off study if intolerable side effects occur.

This is an investigational study. The Food and Drug Administration (FDA) has approved palonosetron and Ondansetron for the prevention of chemotherapy-related nausea and vomiting, and both drugs are commercially available. Up to 150 participants will take part in this study. All will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years with acute myelogenous leukemia or high-risk myelodysplastic syndrome undergoing chemotherapy with high dose cytarabine (1.5 or 2gm/m^2) containing regimens.
2. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

1. Patients with emesis or grade 2 nausea (oral intake is significantly decreased) or 3 nausea (no significant intake requiring intravenous fluids)</= 24 hours before chemotherapy.
2. Patients with ongoing emesis due to any organic etiology.
3. Patients with known hypersensitivity to the study drug or to other selective 5-HT3 receptor antagonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 9/13/2005 to 9/22/2009. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 150 enrolled, only 143 patients were evaluable. Two patients were transferred to intensive care unit, two patients did not receive chemotherapy. One patient received one dose and was placed on hold. One patient received two antiemetic drugs; and 1 patient had a severe headache after two doses and was withdrawn.
Groups:
- Ondansetron: Standard of Care: Standard of care, Ondansetron 8 mg intravenous (IV) as bolus followed by 24 mg IV from 30 minutes before chemotherapy until 12 hours after chemotherapy ends.
- Palonosetron Group 1 (5 Days): Palonosetron once a day 0.25 mg IV injection for 5 days, given over 30 seconds, 30 minutes before chemotherapy.
- Palonosetron Group 2 (3 Days): Palonosetron once a day 0.25 mg IV injection on Days 1, 3, and 5 of chemotherapy, given over 30 seconds, 30 minutes before chemotherapy.
Period: Overall Study
Arm/Group | Ondansetron: Standard of Care | Palonosetron Group 1 (5 Days) | Palonosetron Group 2 (3 Days)
Started | 49 (2 patients were not evaluable in arm 1.) | 51 (3 patients were not evaluable in arm 2) | 50 (2 patients were not evaluable in arm 3.)
Completed | 47 | 48 | 48
Not Completed | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron: Standard of Care | Palonosetron Group 1 (5 Days) | Palonosetron Group 2 (3 Days) | Total
Number analyzed (Participants) | 49 | 51 | 50 | 150
Age Continuous [Median (Full Range); unit: years] | 54 [23 to 69] | 52 [25 to 68] | 53 [18 to 72] | 53 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 21 | 71
  Male | 24 | 26 | 29 | 79
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response
Description: Number of emesis (vomiting) episodes and no use of rescue medication during the administration of chemotherapy assessed as complete response. Complete response is defined as < or equal to 1 episode of emesis during entire 7-day study period, no use of of rescue medication during the study period, and no more than moderate nausea (Grade 2, National Cancer Institutes (NCI) Common Terminology Criteria (CTC)) during chemotherapy.
Time Frame: 7 days, starting first day of chemotherapy
Population: Analysis was per protocol. Seven patients were excluded from the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Ondansetron: Standard of Care | Palonosetron Group 1 (5 Days) | Palonosetron Group 2 (3 Days)
Number analyzed (Participants) | 47 | 48 | 48
participants | 11 | 15 | 18

ADVERSE EVENTS:
Time Frame: 3 years and 7 months
Arm/Group | Ondansetron: Standard of Care | Palonosetron Group 1 (5 Days) | Palonosetron Group 2 (3 Days)
Serious Adverse Events (participants affected / at risk) | 6/49 | 2/51 | 4/50
Other Adverse Events (participants affected / at risk) | 2/49 | 9/51 | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron: Standard of Care (N=49) | Palonosetron Group 1 (5 Days) (N=51) | Palonosetron Group 2 (3 Days) (N=50)
Death (General disorders) | 2 (2) | 0 (0) | 3 (3) — Death is due to disease progression and is unrelated to study drug
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) — Unrelated to study drug
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) — Unrelated to study drug
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) — Unrelated to study drug
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Infection Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Unrelated to study drug
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — Unrelated to study drug
Alanine Aminotransferase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
Febrile Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron: Standard of Care (N=49) | Palonosetron Group 1 (5 Days) (N=51) | Palonosetron Group 2 (3 Days) (N=50)
constipation (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes